CLINICAL TRIAL: NCT02994056
Title: A Phase 2, Multicenter, Open-Label Study to Evaluate the Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed-Dose Combination and Ribavirin for 12 Weeks in Subjects With Chronic HCV Infection and Child-Pugh-Turcotte Class C Cirrhosis
Brief Title: Evaluate the Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed-Dose Combination and Ribavirin for 12 Weeks in Participants With Chronic HCV Infection and Child-Pugh-Turcotte Class C Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-4022; 2016-003066-10 (EudraCT Number)
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2019-09

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SOF/VEL+ RBV (Experimental): SOF/VEL FDC plus RBV for 12 weeks
  Interventions: Drug: SOF/VEL; Drug: RBV

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg FDC tablet administered orally once daily
  Other Names: Epclusa®; GS-7977/GS-5816
Drug: RBV — Tablets administered orally at 600 mg, if well tolerated then up to a maximum total daily dose of 1000 to 1200 mg (based on weight) divided twice daily.

SUMMARY:
The primary objectives of this study are to evaluate the efficacy, safety, and tolerability of the treatment with sofosbuvir velpatasvir (SOF/VEL) fixed-dose combination (FDC) with ribavirin (RBV) for 12 weeks in participants with chronic hepatitis C virus (HCV) infection and Child-Pugh-Turcotte (CPT) Class C cirrhosis.

ELIGIBILITY:
Key Inclusion Criteria:

* A body mass index (BMI) of ≥ 18 kg/m^2
* Chronic HCV infection (≥ 6 months) as documented by either prior medical history or liver biopsy
* Quantifiable HCV RNA at screening
* Individuals may be non-transplanted or with recurrent HCV post-liver transplant.

  * If listed for liver transplant, then the projected date of transplant must be ≥12 weeks after Day1 of treatment
  * If post-liver transplant, then Day1 must be ≥ 6 months from date of transplant
* CPT score of 10 to 12, inclusive, as determined at screening
* Liver imaging within 6 months of Day 1 to exclude hepatocellular carcinoma (HCC)
* If treatment-experienced, the most recent HCV treatment must have been completed at least 8 weeks prior to Screening
* Females of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day 1 prior to randomization
* Males and females of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
* Females must agree to refrain from egg donation and in vitro fertilization during treatment until at least 30 days after the last dose of SOF/VEL or 6 months after the last dose of RBV, whichever occurs last
* Lactating females must agree to discontinue nursing before the study drugs are administered
* Males must agree to refrain from sperm donation from the date of screening until at least 7 months after the last dose of RBV or 30 days after the last dose of SOF/VEL, whichever occurs last
* Adults must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments

Key Exclusion Criteria:

* Current or prior history of any of the following:

  * Clinically significant medical or psychiatric illness or individual is currently under evaluation for a potentially clinically significant illness
  * Gastrointestinal disorder or post-operative condition that could interfere with the absorption of the study drug
  * Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy
  * Significant pulmonary disease, significant cardiac disease or porphyria
  * Malignancy within the 5 years prior to screening, with the exception of specific cancers that have been cured by surgical resection (basal cell skin cancer, etc.). Adults under evaluation for possible malignancy are not eligible
  * Significant drug allergy (such as anaphylaxis or hepatotoxicity)
* Any history of organ transplant other than liver or kidney
* Chronic liver disease of a non-HCV etiology
* Inability to exclude HCC by imaging within 6 months of Day 1
* Alpha-fetoprotein (AFP) > 50 unless negative imaging for hepatic masses within the last 6 months or during screening
* Active spontaneous bacterial peritonitis at screening
* Infection requiring systemic antibiotics at the time of screening
* Evidence of fibrosing cholestatic hepatitis at screening
* Life threatening serious adverse event (SAE) during screening
* Active variceal bleeding within 6 months of screening
* Prior placement of a portosystemic shunt (such as TIPS)
* ECG with clinically significant abnormalities
* Laboratory parameters with clinically significant abnormalities
* Hepatitis B surface antigen positive at screening
* Infection with human immunodeficiency virus (HIV)
* Clinically-relevant alcohol or drug abuse within 12 months of screening. A positive drug screen will exclude individuals unless it can be explained by a prescribed medication; the diagnosis and prescription must be approved by the Investigator
* Prior exposure to any HCV Non-structural Protein 5A (NS5A) inhibitor
* Current use of corticosteroids at any dose >10 mg of prednisone/day (or equivalent dose of corticosteroid)
* Use of any prohibited concomitant medications
* Use of granulocyte macrophage colony-stimulating factor (GM-CSF), epoetin alfa or other hematopoietic stimulating agents within 2 weeks of screening
* Male with pregnant female partner
* History of clinically significant hemoglobinopathy (eg, sickle cell disease, thalassemia)
* Contraindications to RBV therapy
* Known hypersensitivity to VEL, RBV, SOF, the metabolites, or formulation excipients
* Participation in a clinical study with an investigational drug or biologic within 3 months prior to Day 1

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (12):
- United States (10):
  - Tampa General Medical Group, Tampa, Florida
  - Northwestern Memorial Hospital; Clinical Research Unit, Chicago, Illinois
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Southern Therapy and Advanced Research LLC, Jackson, Mississippi
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas
  - Intermountain Liver Disease and Transplant Center, Murray, Utah
  - Bon Secours St. Mary's Hospital of Richmond, Inc. d/b/a Bon Secours Liver Institute of Virginia, Richmond, Virginia
  - University of Washington/ Harborview Medical Center, Seattle, Washington
- France (2):
  - Hopital Henri Mondor, Créteil
  - Hopital Paul Brousse, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Flamm S, Lawitz E, Borg B, Charlton M, Landis C, Reddy R, et al. High Efficacy and Improvement in CPT Class With Sofosbuvir/Velpatasvir Plus Ribavirin for 12 Weeks in Patients With CPT C Decompensated Cirrhosis [Poster THU-138]. EASL: The International Liver Congress; 2019 10-14 April; Vienna, Austria.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States and France. The first participant was screened on 23 January 2017. The last study visit occurred on 12 December 2018.
Pre-assignment Details: 73 participants were screened.
Groups:
- SOF/VEL+ RBV: Sofosbuvir/velpatasvir (SOF/VEL) (400/100 mg) fixed-dose combination (FDC) tablet once daily + ribavirin (RBV) tablet (600-1200 mg based on weight) divided twice daily for 12 weeks in participants with HCV infection and Child-Pugh-Turcotte (CPT) Class C cirrhosis
Period: Overall Study
Arm/Group | SOF/VEL+ RBV
Started | 32
Completed | 23
Not Completed | 9
Not completed — Death | 8
Not completed — Withdrew Consent | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- SOF/VEL+ RBV: SOF/VEL (400/100 mg) FDC tablet once daily + RBV tablet (600-1200 mg based on weight) divided twice daily for 12 weeks in participants with HCV infection and CPT Class C cirrhosis
Arm/Group | SOF/VEL+ RBV
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Black or African American Native | 6
  White | 18
  Not Permitted | 6
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 26
  France | 6
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.2 (1.19)
HCV RNA Category [Count of Participants; unit: Participants]
  < 800,000 IU/mL | 23
  ≥ 800,000 IU/mL | 9
IL28B [Count of Participants; unit: Participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  Participants
    CC | 15
    CT | 14
    TT | 3
Child-Pugh-Turcotte Class [Count of Participants; unit: Participants] — CPT is a chronic liver disease classification system. Classes include CPT Class A, CPT Class B, and CPT Class C, in order of greater disease severity.
  Participants
    CPT B [7-9] | 9
    CPT C [10-15] | 23
Model for End Stage Liver Disease (MELD) Score Category [Count of Participants; unit: Participants] — MELD score is a chronic liver disease severity scoring system. Scores can range from 6 to 40, with higher scores indicating greater disease severity.
  Participants
    10-15 MELD Score | 13
    16-20 MELD Score | 17
    21-25 MELD Score | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: The Full Analysis Set included all enrolled participants who took at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOF/VEL+ RBV (Total): SOF/VEL (400/100 mg) FDC tablet once daily + RBV tablet (600-1200 mg based on weight) divided twice daily for 12 weeks in participants with HCV infection and CPT Class C cirrhosis
- SOF/VEL+ RBV (GT-1): SOF/VEL (400/100 mg) FDC tablet once daily + RBV tablet (600-1200 mg based on weight) divided twice daily for 12 weeks in participants with genotype 1 (GT-1) HCV infection and CPT Class C cirrhosis
- SOF/VEL+ RBV (GT-2): SOF/VEL (400/100 mg) FDC tablet once daily + RBV tablet (600-1200 mg based on weight) divided twice daily for 12 weeks in participants with genotype 2 (GT-2) HCV infection and CPT Class C cirrhosis
- SOF/VEL+ RBV (GT-3): SOF/VEL (400/100 mg) FDC tablet once daily + RBV tablet (600-1200 mg based on weight) divided twice daily for 12 weeks in participants with genotype 3 (GT-3) HCV infection and CPT Class C cirrhosis
Arm/Group | SOF/VEL+ RBV (Total) | SOF/VEL+ RBV (GT-1) | SOF/VEL+ RBV (GT-2) | SOF/VEL+ RBV (GT-3)
Number analyzed (Participants) | 32 | 18 | 5 | 7
percentage of participants | 78.1 [60.0 to 90.7] | 72.2 [46.5 to 90.3] | 80.0 [28.4 to 99.5] | 85.7 [42.1 to 99.6]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Study Drug (SOF/VEL or RBV) Due to an Adverse Event
Time Frame: First dose date up to Week 12
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL+ RBV
Number analyzed (Participants) | 32
percentage of participants
  Discontinuation of SOF/VEL | 6.3
  Discontinuation of RBV | 21.9

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 4 Weeks After Discontinuation of Therapy (SVR4)
Description: SVR4 was defined as HCV RNA < LLOQ 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- SOF/VEL+ RBV (Total): SOF/VEL (400/100 mg) FDC tablet once daily + ribavirin RBV tablet (600-1200 mg based on weight) divided twice daily for 12 weeks in participants with HCV infection and CPT Class C cirrhosis
Arm/Group | SOF/VEL+ RBV (Total) | SOF/VEL+ RBV (GT-1) | SOF/VEL+ RBV (GT-2) | SOF/VEL+ RBV (GT-3)
Number analyzed (Participants) | 32 | 18 | 5 | 7
percentage of participants | 87.5 [71.0 to 96.5] | 88.9 [65.3 to 98.6] | 80.0 [28.4 to 99.5] | 85.7 [42.1 to 99.6]

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 24 Weeks After Discontinuation of Therapy (SVR24)
Description: SVR24 was defined as HCV RNA < LLOQ at 24 weeks after stopping study treatment.
Time Frame: Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL+ RBV (Total) | SOF/VEL+ RBV (GT-1) | SOF/VEL+ RBV (GT-2) | SOF/VEL+ RBV (GT-3)
Number analyzed (Participants) | 32 | 18 | 5 | 7
percentage of participants | 75.0 [56.6 to 88.5] | 72.2 [46.5 to 90.3] | 80.0 [28.4 to 99.5] | 71.4 [29.0 to 96.3]

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ While on Study Treatment
Time Frame: Weeks 2, 4, 8, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SOF/VEL+ RBV (Total) | SOF/VEL+ RBV (GT-1) | SOF/VEL+ RBV (GT-2) | SOF/VEL+ RBV (GT-3)
Number analyzed (Participants) | 32 | 18 | 5 | 7
Percentage of participants
  Week 2 | 43.8 [26.4 to 62.3] | 38.9 [17.3 to 64.3] | 0 [0.0 to 52.2] | 71.4 [29.0 to 96.3]
  Week 4: number analyzed (Participants) | 29 | 16 | 4 | 7
  Week 4 | 96.6 [82.2 to 99.9] | 100.0 [79.4 to 100.0] | 75.0 [19.4 to 99.4] | 100.0 [59.0 to 100.0]
  Week 8: number analyzed (Participants) | 29 | 16 | 4 | 7
  Week 8 | 100.0 [88.1 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [59.0 to 100.0]
  Week 12: number analyzed (Participants) | 29 | 16 | 4 | 7
  Week 12 | 100.0 [88.1 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [39.8 to 100.0] | 100.0 [59.0 to 100.0]

6. Secondary Outcome: Percentage of Participants With No Change, Improved, and Worsened Child-Pugh-Turcotte (CPT) Class
Description: CPT is a chronic liver disease classification system. Classes include CPT Class A, CPT Class B, and CPT Class C, in order of greater disease severity. Participants with improved CPT class was defined as having Class C at Baseline and Class B or A at Posttreatment Week 24 or Class B at Baseline and Class A at Posttreatment Week 24. Participants with worsened CPT class was defined as having Class A at Baseline and Class B or C at Posttreatment Week 24 or Class B at Baseline and Class C at Posttreatment Week 24. Participants with no change CPT class was defined as having CPT Class same between Baseline and Posttreatment Week 24.
Time Frame: Baseline to Posttreatment Week 24
Population: Participants in the Full Analysis Set who achieved SVR24 with available data were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | SOF/VEL+ RBV
Number analyzed (Participants) | 19
Percentage of participants
  Improved CPT Class | 42.1
  Worsened CPT Class | 0
  No Change CPT Class | 57.9

7. Secondary Outcome: Percentage of Participants With a Decrease, No Change, or Increase in Model for End Stage Liver Disease (MELD) Score
Description: MELD score is a chronic liver disease severity scoring system. Scores can range from 6 to 40, with higher scores indicating greater disease severity. "No change" was assigned for differences (posttreatment visits minus baseline score) of -1, 0 or 1; "Decrease" was assigned for differences that were less than or equal to -2; and "Increase" was assigned for values that were greater than or equal to 2.
Time Frame: Baseline to Posttreatment Week 24
Population: Participants in the Full Analysis Set who achieved SVR24 with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL+ RBV
Number analyzed (Participants) | 19
percentage of participants
  Decrease (Improvement) | 52.6
  No Change | 21.1
  Increase (Worsening) | 26.3

8. Secondary Outcome: Absolute HCV RNA Level Through Week 12
Time Frame: Baseline; Weeks 2, 4, 8, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+ RBV (Total) | SOF/VEL+ RBV (GT-1) | SOF/VEL+ RBV (GT-2) | SOF/VEL+ RBV (GT-3)
Number analyzed (Participants) | 32 | 18 | 5 | 7
log10 IU/mL
  Baseline | 5.17 (1.187) | 5.46 (0.537) | 6.01 (0.502) | 4.84 (1.058)
  Week 2: number analyzed (Participants) | 29 | 16 | 4 | 7
  Week 2 | 1.46 (0.392) | 1.47 (0.387) | 1.63 (0.150) | 1.43 (0.526)
  Week 4: number analyzed (Participants) | 28 | 16 | 3 | 7
  Week 4 | 1.15 (0.00) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000)
  Week 8: number analyzed (Participants) | 29 | 16 | 4 | 7
  Week 8 | 1.15 (0.00) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000)
  Week 12: number analyzed (Participants) | 29 | 16 | 4 | 7
  Week 12 | 1.15 (0.00) | 1.15 (0.000) | 1.15 (0.000) | 1.15 (0.000)

9. Secondary Outcome: Change From Baseline in HCV RNA
Time Frame: Baseline; Weeks 2, 4, 8, and 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL+ RBV (Total) | SOF/VEL+ RBV (GT-1) | SOF/VEL+ RBV (GT-2) | SOF/VEL+ RBV (GT-3)
Number analyzed (Participants) | 29 | 16 | 4 | 7
log10 IU/mL
  Change at Week 2 | -3.72 (1.092) | -4.06 (0.531) | -4.50 (0.366) | -3.41 (0.665)
  Change at Week 4: number analyzed (Participants) | 28 | 16 | 3 | 7
  Change at Week 4 | -3.99 (1.238) | -4.39 (0.520) | -4.88 (0.395) | -3.70 (1.058)
  Change at Week 8 | -4.00 (1.217) | -4.39 (0.520) | -4.72 (0.445) | -3.70 (1.058)
  Change at Week 12 | -4.00 (1.217) | -4.39 (0.520) | -4.72 (0.445) | -3.70 (1.058)

10. Secondary Outcome: Number of Participants With Virologic Failure
Description: Virologic failure was defined as:
  * On-treatment virologic failure:
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  * Virologic relapse:
    * Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit
Time Frame: Baseline up to Posttreatment Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | SOF/VEL+ RBV (GT-1) | SOF/VEL+ RBV (GT-2) | SOF/VEL+ RBV (GT-3) | SOF/VEL+ RBV (Total)
Number analyzed (Participants) | 18 | 5 | 7 | 32
Participants | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to Week 12 plus 30 days; All-Cause Mortality: First dose date up to Posttreatment Week 24
Description: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | SOF/VEL+ RBV
All-Cause Mortality (participants affected / at risk) | 8/32
Serious Adverse Events (participants affected / at risk) | 17/32
Other Adverse Events (participants affected / at risk) | 27/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL+ RBV (N=32)
Atrial fibrillation (Cardiac disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Dermo-hypodermitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Mixed hepatocellular cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL+ RBV (N=32)
Anaemia (Blood and lymphatic system disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 5
Asthenia (General disorders) | 6
Fatigue (General disorders) | 2
Oedema peripheral (General disorders) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 2
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2016-11-22): https://cdn.clinicaltrials.gov/large-docs/56/NCT02994056/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT02994056/SAP_001.pdf